CLINICAL TRIAL: NCT02822989
Title: Using the Cholinergic Anit-Inflammatory Pathway to Treat Systemic Lupus Musculoskeletal Pain
Brief Title: Using the Cholinergic Anti-Inflammatory Pathway to Treat Systemic Lupus Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Northwell Health (Other)
Collaborators: John and Marcia Goldman Foundation (Unknown)
Responsible Party: Principal Investigator, Cynthia Aranow, MD, Investigator, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0171
Record Dates: First submitted 2016-05-26; First posted 2016-07-06 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Lupus Erythematosus, Systemic; Musculoskeletal Pain
Keywords: Lupus Erythematosus, Systemic; Musculoskeletal Pain; Inflammation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Musculoskeletal Pain; Inflammation | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Stimulation (Active Comparator): Subjects randomized to this arm will receive transcutaneous vagus nerve stimulation for 5 minutes on 4 consecutive days.
  Interventions: Device: Vagus nerve stimulation
- Sham Vagus Nerve Stimulation (Sham Comparator): Subjects randomized to this arm will receive sham stimulation for 5 minutes for 4 consecutive days.
  Interventions: Device: Sham vagus nerve stimulation

INTERVENTIONS:
Device: Vagus nerve stimulation — Patients will receive transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes daily for 4 consecutive days. The device is a handheld electrical pulse generator and a pair of electrodes to be placed at the ear for stimulation. The specific target at the ear will be the auricular branch of the vagus nerve which innervates the skin of the ear canal. Electrodes will be placed near/at the entrance to the canal of the ear to provide stimulation to the auricular branch.
  Arms: Vagus Nerve Stimulation
Device: Sham vagus nerve stimulation — Patients will receive sham transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes daily for 4 consecutive days. Sham stimulation will be performed in the identical manner as true transcutaneous stimulation except that the patient will not receive electrical stimulation of the vagus nerve.
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune, inflammatory disease and musculoskeletal pain is one of the most common symptoms. This study will investigate whether transcutaneous stimulation of the vagus nerve will decrease lupus musculoskeletal pain. This study will additionally investigate the biologic effects of vagus nerve stimulation on inflammation. It will be the first clinical study using one of the body's own pathways of modulating the immune system and inflammatory response, the cholinergic anti-inflammatory pathway, in SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. SLE (defined by the ACR or SLICC criteria),
3. Musculoskeletal pain ≥ 4 on a non-anchored VAS 10 cm scale
4. BILAG C on Musculoskeletal Domain of the BILAG 2004
5. If on corticosteroids, the dose must be stable and ≤ 10mg/day (prednisone or equivalent) for at least 28 days before baseline,
6. If on background immunosuppressive treatment the dose must be stable for at least 28 days before baseline
7. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Treatment with rituximab within one year of baseline (subjects with previous treatment with rituximab can enter study only with documentation of B cell repletion),
2. Treatment with cyclophosphamide within 2 months of baseline,
3. Expectation to increase steroids and/or immunosuppressive treatment,
4. Anti-phospholipid syndrome,
5. Fibromyalgia (fibromyalgia will be defined as a score > 13 on the Fibromyalgia Symptom Scale (FSS).
6. Treatment with an anti-cholinergic medication, including over the counter medications,
7. Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
8. Current tobacco or nicotine user,
9. Joint replacement within 60 days prior to study enrollment or planned within the course of the study,
10. Any planned surgical procedure requiring general anesthesia within the course of the study,
11. Intra-articular cortisone injections within 28 days of the start of study,
12. Chronic inflammatory disorders apart from SLE affecting the joints,
13. Investigational drug and/or treatment during the 28 days or seven half-lives of the investigational drug prior to the start of study drug dosing (Day 0), whichever is the greater length of time,
14. Active infection including hepatitis B or hepatitis C at baseline,
15. Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention,
16. Pregnancy or lactation,
17. Comorbid disease that may require administration of corticosteroid use,
18. Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal pain. | 5 days
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.

SECONDARY OUTCOMES:
SLE Disease activity | 5 days
  SLE disease activity will be assessed using the SLEDAI, a validated disease activity instrument for SLE.
Fatigue | 5 days
  Fatigue will be measured using the FACET F questionnaire which will be completed by each subject.
Fatigue | 12 days
  Fatigue will be measured using the FACET F questionnaire which will be completed by each subject.
Tender and swollen joint counts | 5 days
  The number of tender and swollen joints of the subject will be assessed by the investigator who will examine 68 potential tender joints and 66 potential swollen joints.
Tender and swollen joint counts | 12 days
  The number of tender and swollen joints of the subject will be assessed by the investigator who will examine 68 potential tender joints and 66 potential swollen joints.
SLE cutaneous activity | 5 days
  Cutaneous activity will be assessed using the CLASI, a validated index for SLE skin disease.
SLE cutaneous activity | 12 days
  Cutaneous activity will be assessed using the CLASI, a validated index for SLE skin disease.
Musculoskeletal Pain | 12 days
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.
Percentage of subjects with treatment emergent adverse events. | 12 days
  The percentage of participants with treatment emergent adverse events will be assessed using the NCI-CTAEversion4.

OTHER OUTCOMES:
TNF, HMGB1, IL-6, Il1B, IFNα and IL10 levels | 5 days
  Levels of inflammatory cytokines (ie TNF, HMGB1, IL-6, Il1B, IFNα and IL10) will be measured in patients sera.
TNF, HMGB1, IL-6, Il1B, IFNα and IL10 levels | 12 days
  Levels of inflammatory cytokines (ie TNF, HMGB1, IL-6, Il1B, IFNα and IL10) will be measured in patients sera.
Lipopolysaccharide stimulated levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 in whole blood. | 5 days
  Whole blood will be taken from patients and stimulated by lipopolysaccharide. Levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 that are produced by the cells in the whole blood will be measured.
Lipopolysaccharide stimulated levels of TNF, IL-6, Il1B, IFNα and IL10 in whole blood. | 12 days
  Whole blood will be taken from patients and stimulated by lipopolysaccharide. Levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 that are produced by the cells in the whole blood will be measured.
Gardiquimod stimulated levels of TNF, IL-6, Il1B, IFNα and IL10 in whole blood. | 5 days
  Whole blood will be taken from patients and stimulated by gardiquimod.. Levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 that are produced by the cells in the whole blood will be measured.
Gardiquimod stimulated levels of TNF, IL-6, Il1B, IFNα and IL10 in whole blood. | 12 days
  Whole blood will be taken from patients and stimulated by gardiquimod.. Levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 that are produced by the cells in the whole blood will be measured.
CpG stimulated levels of TNF, IL-6, Il1B, IFNα and IL10 in whole blood. | 5 days
  Whole blood will be taken from patients and stimulated by CpG. Levels of TNF, HMGB1, IL-6, Il1B, IFNα and IL10 that are produced by the cells in the whole blood will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, M.D., Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069